CLINICAL TRIAL: NCT03072433
Title: The Effect of an Intervention Program for Primary Caregivers on the Development of Children With Severe Malnutrition: A Cluster Randomized Controlled Clinical Trial
Brief Title: An Intervention for Primary Caregivers to Improve Outcomes in Children With Severe Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Principal Investigator, Robert Bandsma, Staff Gastroenterologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1000053078
Record Dates: First submitted 2017-02-17; First posted 2017-03-07 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Child Malnutrition
Keywords: child malnutrition; child development; counseling
MeSH Terms: conditions — Child Nutrition Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Comparison group will receive the current standard of care. Nurses are instructed to tell mothers about nutrition and water, sanitation and hygiene at any point prior to discharge from hospital. In addition, nurses will tell primary caregivers to play with their children even while they are receiving treatment in a play area with toys available.
  Interventions: Behavioral: Standard of Care
- Counseling Intervention Package (Experimental): Primary caregivers in the intervention group receive group education sessions involving psychosocial stimulation, nutrition and feeding, and water, sanitation and hygiene components during a total of four days.
  Interventions: Behavioral: Counseling Intervention Package

INTERVENTIONS:
Behavioral: Counseling Intervention Package — Daily 45 minutes of group teaching for primary caregivers, followed by 45 minutes of supervised play and stimulation with their children for a total of four days. Teaching modules consist of psychosocial stimulation, nutrition and feeding, and water, sanitation and hygiene practices.
  Other Names: Kusamala Program
  Arms: Counseling Intervention Package
Behavioral: Standard of Care — Nutrition and water sanitation and hygiene counseling at any point prior to discharge from hospital as per the local nutrition rehabilitation unit standard of care. In addition, primary caregivers will be stimulated to play with their children in a play area.
  Arms: Standard of Care

SUMMARY:
This cluster-randomized controlled trial will evaluate the effectiveness of a four-day hospital-based intervention program for primary caregivers of children with severe malnutrition.

DETAILED DESCRIPTION:
Mortality rates remain high in hospitalized children with severe malnutrition and long-term impairments in child development exist in children that do survive. Hospitalized children with severe malnutrition will be allocated to an intervention or standard of care group in each one-week cycle. The intervention package consists of a counseling and support program that includes three modules: 1) psychosocial stimulation; 2) nutrition and feeding; and 3) water, sanitation and hygiene. Assessments will be done at baseline (t=0) and follow-up (t=6 months). The primary outcome is child development, which will be assessed using the Malawi Developmental Assessment Tool, a validated tool for gross and fine motor, language, and social development.

ELIGIBILITY:
Inclusion Criteria:

* Child 6-59 months of age with severe malnutrition
* Child admitted to hospital because of severe malnutritionwith medical complications as defined by the current World Health Organization guidelines or has no appetite if there are no complications
* Primary caregiver (self-identified) present at hospital.

Exclusion Criteria:

* Primary caregiver declined to give informed consent;
* Child with a known terminal illness (i.e. in the opinion of the treating physician the child is likely to die within six months)
* Child requires a surgical procedure.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Malawi Developmental Assessment Tool Score | 6 months post-discharge from hospital
  Gross motor, fine motor, language, and social development

SECONDARY OUTCOMES:
Nutritional status based on: mid-upper arm circumference (MUAC) | 6 months post-discharge from hospital
  MUAC in millimeters
Nutritional status based on: World Health Organization (WHO) z-scores | 6 months post-discharge from hospital
  Weight-for-length or -height z-scores and height-for-age z-scores
Nutritional status based on: nutritionally-induced bilateral pitting oedema | 6 months post-discharge from hospital
  Bilateral pitting oedema
Duration of hospital stay | During hospitalization; up to three days before enrollment until discharge from hospital (e.g., up to 30 days)
  Number of days that hospital treatment is required
Appetite | During hospitalization; up to three days before enrollment until discharge from hospital (e.g., up to 30 days)
  Number of days that nasogastric tube is required
Clinical deterioration | During hospitalization; up to three days before enrollment until discharge from hospital (e.g., up to 30 days)
  Number of clinical danger signs
Readmission | Within 6 months post-discharge from hospital
  Requiring inpatient treatment
Mortality | Within 6 months post-discharge from hospital
  Inpatient or post-discharge mortality

OTHER OUTCOMES:
Self Reporting Questionnaire (SRQ-20) | 6 months post-discharge from hospital
  Mental health of primary caregivers
Home Observation for Measurement of the Environment (HOME) Inventory | 6 months post-discharge from hospital
  Stimulus and support for children in the household
Primary caregiver knowledge, attitudes, and practices | 6 months post-discharge from hospital
  Questionnaire with the following modules: hygiene and sanitation, nutrition and feeding with a 24-hour food recall of the child (follow-up only), and malnutrition knowledge and attitudes
Participant engagement | Day one of the intervention during hospital stay
  Attendance of participants on day one of the intervention program
Participant adherence | Across the four days of the intervention during hospital stay
  Attendance of participants on all four days of the intervention program

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bandsma, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniel AI, Bwanali M, Tenthani JC, Gladstone M, Voskuijl W, Potani I, Ziwoya F, Chidzalo K, Mbale E, Heath A, Bourdon C, Njirammadzi J, van den Heuvel M, Bandsma RHJ. A Mixed-Methods Cluster-Randomized Controlled Trial of a Hospital-Based Psychosocial Stimulation and Counseling Program for Caregivers and Children with Severe Acute Malnutrition. Curr Dev Nutr. 2021 Jul 21;5(8):nzab100. doi: 10.1093/cdn/nzab100. eCollection 2021 Aug. PMID 34447897
- [Derived] Daniel AI, van den Heuvel M, Gladstone M, Bwanali M, Voskuijl W, Bourdon C, Potani I, Fernandes S, Njirammadzi J, Bandsma RHJ. A mixed methods feasibility study of the Kusamala Program at a nutritional rehabilitation unit in Malawi. Pilot Feasibility Stud. 2018 Sep 24;4:151. doi: 10.1186/s40814-018-0347-8. eCollection 2018. PMID 30258650
- [Derived] Daniel AI, van den Heuvel M, Voskuijl WP, Gladstone M, Bwanali M, Potani I, Bourdon C, Njirammadzi J, Bandsma RHJ. The Kusamala Program for primary caregivers of children 6-59 months of age hospitalized with severe acute malnutrition in Malawi: study protocol for a cluster-randomized controlled trial. Trials. 2017 Nov 17;18(1):550. doi: 10.1186/s13063-017-2299-3. PMID 29149905